CLINICAL TRIAL: NCT07231107
Title: Comparative Study Between Airway Pressure Release Ventilation and Pressure Regulated Volume Control (PRVC) in Protective Lung Strategy as a Recruitment Maneuver for Severe ARDS Mechanically Ventilated Patients Using Lung Ultrasound Score
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed Shaban, post graduate student, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: FMASU MD 190/2022
Record Dates: First submitted 2025-09-29; First posted 2025-11-17 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: ARDS (Acute Respiratory Distress Syndrome)
Keywords: Lung ultrasound; APRV; recruitment
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRVC ventilated ARDS patients (Active Comparator): managed by using conventional lung protective strategy using Pressure regulated volume control mode (PRVC) and positive end expiratory pressure, initial setting Tidal volume (VT):4-6ml/kg predicted body weight, PEEP according to ARDSnet guidelines recommendation for Low tidal volume high strategy.
  Interventions: Procedure: Lung ultrasound
- APRV ventilated ARDS patients (Active Comparator): managed by airway pressure release ventilation mode initial settings Phigh:25 Plow:0 Thigh: 4.5 Tlow: 0.5 Fio2: 1. Options for setting the Phigh either premeasured Pplat or according to the Oxygenation index.
  Interventions: Procedure: Lung ultrasound

INTERVENTIONS:
Procedure: Lung ultrasound — bedside lung ultrasound in six lung regions of interest, delineated by a parasternal line, anterior axillary line, posterior axillary line, and paravertebral line, are examined on each side. Each lung region is carefully examined in the longitudinal plane, and each intercostal space present in the region is examined in the transversal plane. The worst ultrasound pattern characterizes the region (regional LUS) using the following grading: 0 = normal aeration; 1 = moderate loss of aeration (interstitial syndrome, defined by multiple spaced B lines, or localized pulmonary edema, defined by coalescent B lines in less than 50% of the intercostal space examined in the transversal plane, or subpleural consolidations); 2 = severe loss of aeration (alveolar edema, defined by diffused coalescent B lines occupying the whole intercostal space); and 3 = complete loss of lung aeration (lung consolidation defined as a tissue pattern with or without air bronchogram)

SUMMARY:
The aim of this study is to elaborate on the effectiveness of recruitment maneuver by airway pressure release ventilation (APRV) as an open lung ventilatory strategy in comparison with PRVC mode in lung protective strategy regarding improvement of LUS score and P/F ratio in patients with severe ARDS

DETAILED DESCRIPTION:
Acute Respiratory distress syndrome (ARDS) is the most severe form of acute lung injury (ALI) which still has high rates of morbidity and mortality. Mechanical ventilation is still the backbone of patient management. One of the newly developed and successfully used strategies in patients with ARDS is lung protective strategies (LPS). However, use of low tidal volumes during LPS may be associated with atelectasis due to decreased alveolar inflation.

In acute respiratory distress syndrome (ARDS) patients, a recruitment strategy combines recruitment maneuvers (RMs) and positive end-expiratory pressure (PEEP) to prevent atelectrauma. Recruitment maneuvers are a voluntary strategy for effecting a temporary increase in trans-pulmonary pressure (PL), which in turn should reopen those alveolar units that are either poorly aerated or not aerated at all. PEEP may decrease ventilator-induced lung injury (VILI) by keeping those lung regions open that may otherwise collapse The Open lung approach is another ventilatory strategy complementary with the concept of protective ventilation. Lachmann was the first who introduced the open lung concept combining a lung recruitment maneuver (RM) with a sufficient level of PEEP. Recruitment maneuvers minimize the impact of the two known VILI mediators: tidal over distension (i.e., alveoli that receive volume and pressure that exceed their elastic limit) and tidal recruitment (i.e., the repetitive opening and closing of atelectasis during mechanical breathing), Airway pressure release ventilation (APRV) is one of the newly introduced modes in ARDS management. It is a pressure-controlled mode that uses two levels of pressures with inverted ratio ventilation. Release of airway pressure during APRV simulates expiration while elevated baseline pressure improves oxygenation. One of the advantages of this mode is that it allows spontaneous breathing It is considered an alternative, life-saving modality in patients with acute respiratory distress syndrome (ARDS) who struggle for oxygenation. Compared to the classical ventilation, APRV has been shown to provide lower peak pressure, better oxygenation, less circulatory loss, and better gas exchange without deteriorating the hemodynamic condition of the ARDS patient. This mode is believed to help to achieve the target of opening consolidated lung areas (recruitment) and to prevent repeated opening-closing of alveoli (recruitment). However, there still needs to be more and more proof to support this hypothesis. Recently, it has been proposed that the early use of protective mechanical ventilation with APRV could be used preemptively to prevent the development of ARDS in high-risk patients Lung Ultrasound has favorable features to assess RM due to its high specificity and sensitivity to detect lung collapse together with its non-invasiveness, availability, and simple use at the bedside. Ultrasound also has the capability of providing a differential diagnosis between atelectasis and lung consolidation of other origin such as pneumonia. The bilateral distribution of consolidations, presence of static air bronchograms, images of tidal recruitment within consolidation and absence of a companion pleural effusion strongly support the diagnosis of atelectasis. Furthermore, retrospectively the disappearance of the lung consolidation pattern after a RM confirms the diagnosis Acute respiratory distress syndrome (ARDS) is a severe life-threatening lung reaction to various forms of injuries that cause hypoxia. it has been demonstrated that mechanical ventilation by lung protection strategy can be provided in patients with ARDS, resulting in better pulmonary function and higher rates of weaning from the ventilator. lung-protective strategy was associated with improved survival in 28 days and a lower rate of barotrauma in patients with acute respiratory distress syndrome. Protective ventilation was not associated with a higher rate of survival to hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-60 years old.
* Sex: both males and females
* Accepts health volunteers: No
* all Patients who were mechanically ventilated and diagnosed to have ARDS due to sepsis according to Berlin definition.

During the course of the study, a new global definition for ARDS was introduced. To ensure our findings align with the most updated classification, we modified our inclusion criteria to incorporate the new global definition. Patients meeting the Berlin Definition or the new definition were included.

Berlin Definition of the acute respiratory distress syndrome (ARDS) Acute Respiratory Distress Syndrome Timing Within 1 week of a known clinical insult or new or worsening respiratory Symptoms Chest imaging Bilateral opacities - not fully explained by effusion, lobar/lung collapse, or nodules. Origin of edema Respiratory failure not fully explained by cardiac failure or fluid overload need objective assessment (eg, echocardiography) to exclude hydrostatic edema if no risk factor present.

Oxygenation Mild 200 mmHg <Pao2/Fio2 < 300 mmHg with PEEP or CPAP > 5 cmH2O. Moderate 100 mmHg <Pao2/Fio2 < 200 mmHg with PEEP > 5 cmH2O. Severe Pao2/Fio2 < 100 mmHg with PEEP > 5 cmH2O. (Gordon D, et al; 2012). Diagnostic Criteria for the New Global Definition of ARDS Acute Respiratory Distress Syndrome Risk factors and origin of edema Precipitated by an acute predisposing risk factor, such as pneumonia, non-pulmonary infection, trauma, transfusion, aspiration, or shock.

Pulmonary edema is not exclusively or primarily attributable to cardiogenic pulmonary edema/fluid overload, and hypoxemia/gas exchange abnormalities are not primarily attributable to atelectasis. However, ARDS can be diagnosed in the presence of these conditions if a predisposing risk factor for ARDS is also present.

Timing Acute onset or worsening of hypoxemic respiratory failure within 1 week of the estimated onset of the predisposing risk factor or new or worsening respiratory symptoms.

Chest imaging Bilateral opacities on chest radiography and computed tomography or bilateral B lines and/or consolidations on ultrasound* not fully explained by effusions, atelectasis, or nodules / masses.

Oxygenation Non-intubated ARDS Intubated ARDS Modified Definition for Resource-Limited Settings

* PaO2:FIO2<300mmHg or
* SpO2:FIO2<315 (if SpO2<97%) on HFNO with flow of >30 L/min or NIV/CPAP with at least 5 cm H2O end-expiratory pressure Mild:
* 200<PaO2:FIO2<300 mm Hg Or
* 235<SpO2:FIO2<315 (if SpO2<97%)

Moderate:

* 100, PaO2:FIO2<200 mm Hg or
* 148<SpO2:FIO2<235 (if SpO2<97%)

Severe:

* PaO2:FIO2<100 mm Hg or
* SpO2:FIO2<148 (if SpO2<97%) • SpO2:FIO2<315 (if SpO2<97%).
* Neither positive end-expiratory pressure nor a minimum flow rate of oxygen is required for diagnosis in resource-limited settings.

(Matthay MA, et al; 2024).

Exclusion Criteria:

* Patient refusal
* Patient with advanced cardiac disorders (rheumatic or ischemic).
* Patients with COPD, pneumothorax, surgical emphysema.
* Patients with advanced liver or renal disorders
* Patients with advanced malignancy.
* Female patients during pregnancy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2022-08-18 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
lung ultrasound score | 7 days started after mechanical ventilation
  assessment of the lung interstitial tissue by ultrasound Ultrasound patterns at different degrees of lung aeration.
  1. Normal lung ultrasound pattern (score = 0).
  2. Well-Spaced B lines (moderate loss of aeration; score = 1).
  3. Coalescent B lines (severe loss of aeration; score = 2).
  4. Consolidated lung (complete loss of aeration; score = 3).
P/F Ratio (Pao2/Fio2 Ratio) | 7 days started after mechanical ventilation
  ratio between the Partial pressure of Oxygen and the fraction of inspired oxygen Mild ARDS: 200 mmHg <Pao2/Fio2 < 300 mmHg Moderate ARDS:100 mmHg <Pao2/Fio2 < 200 mmHg Severe ARDS: Pao2/Fio2 < 100 mmHg

SECONDARY OUTCOMES:
Heart rate. (BPM). | every 24 hours for 7 days after mechanical ventilation
  heart rate in beat per minute
Invasive Mean arterial blood pressure. (mmHG). | every 24 hours for 7 days after mechanical ventilation
  mean arterial blood pressure in mmHg
Vasopressor-Inotrope score (VIS) | every 24 hours for 7 days after mechanical ventilation
  Vasopressor dose monitored daily using Vasopressor-Inotrope score (VIS) calculated as: Vasoactive-Inotropic Score = dopamine dose (µg/kg/min) + dobutamine dose (µg/kg/min) + 100 x adrenaline dose (µg/ kg/ min) + 100 x noradrenaline dose (µg/kg/min) + 10 x milrinone dose (µg/kg/min) + 10.000 x vasopressin dose (U/kg/min)
Lung compliance. (mL/cmH2O). | every 24 hours for 7 days after mechanical ventilation
  Lung compliance. (mL/cmH2O) calculated as change in tidal volume divided by the change in ventilating pressures
Oxygenation index | every 24 hours for 7 days after mechanical ventilation
  Oxygenation index calculated as: mean airway pressure *Fio2*100) /Pao2
Length of stay. (Days) | through study completion, From date of admission until the date of discharge or transfer or date of death from any cause, whichever came first, assessed up to 1 month
  total Length of stay through study completion, From date of admission until the date of discharge or transfer or date of death from any cause, whichever came first, assessed up to 1 month
Total ventilation days | calculated From date of endotracheal intubation until the date of extubation or date of death from any cause, whichever came first, assessed up to 1 month
  calculated from date of endotracheal intubation until the date of extubation or date of death from any cause, whichever came first, assessed up to 1 month
outcome | through study completion, From date of admission until the date of discharge or transfer or date of death from any cause, whichever came first, assessed up to 1 month"
  final outcome of the patient dicharged or improved, transferred or died

OTHER OUTCOMES:
SOFA score | Every 24 hours for 7 day
  Sequential organ failure assessment score for daily assessment of the septic shock patient
LIS score | Every 24 hours for 7 day
  Lung injury score daily assessment LIS, each of the four components is categorized from 0 to 4, where a higher number is worse. The total LIS is obtained by dividing the aggregate sum by the number of components used.
  Chest radiograph score No alveolar consolidation= 0 Alveolar consolidation confined to 1 quadrant= 1 Alveolar consolidation confined to 2 quadrants=2 Alveolar consolidation confined to 3 quadrants= 3 Alveolar consolidation in all 4 quadrants= 4 Hypoxemia score PaO2/FIO2: ≥ 300= 0 PaO2/FIO2: 225 to 299=1 PaO2/FIO2: 175 to 224= 2 PaO2/FIO2: 100 to 174= 3 PaO2/FIO2: <100= 4 PEEP score (when ventilated) PEEP: ≤ 5 cm H2O= 0 PEEP: 6 to 8 cm H2O= 1 PEEP: 9 to 11 cm H2O= 2 PEEP: 12 to 14 cm H2O= 3 PEEP: ≥ 15 cm H2O= 4 Respiratory system compliance score Compliance: ≥ 80 ml/cm H2O= 0 Compliance: 60 to 79 ml/cm H2O= 1 Compliance: 40 to 59 ml/cm H2O= 2 Compliance: 20 to 39 ml/cm H2O= 3 Compliance: ≤19 ml/cm H2O= 4
Mean airway pressure (Paw) | Every 24 hours for 7 day
  Paw = 0.5 X (PIP - PEEP) X (TI/Ttot) + PEEP
Airway Resistance | Every 24 hours for 7 day
  Airway resistance calculated as [(ppeak-pplat)/(flow/60)]
Mechanical power | Every 24 hours for 7 day
  Mechanical power calculated as [0.098*Vt*RR*(Ppeak-0.5 ∆ pressure)]/1000 less than 17 is lung protective strategy

CONTACTS AND LOCATIONS:
Locations (1):
- Ainshams University, Cairo, Abbasia, Egypt

REFERENCES:
- [Result] ARDS Definition Task Force; Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: the Berlin Definition. JAMA. 2012 Jun 20;307(23):2526-33. doi: 10.1001/jama.2012.5669. PMID 22797452
- [Result] Matthay MA, Arabi Y, Arroliga AC, Bernard G, Bersten AD, Brochard LJ, Calfee CS, Combes A, Daniel BM, Ferguson ND, Gong MN, Gotts JE, Herridge MS, Laffey JG, Liu KD, Machado FR, Martin TR, McAuley DF, Mercat A, Moss M, Mularski RA, Pesenti A, Qiu H, Ramakrishnan N, Ranieri VM, Riviello ED, Rubin E, Slutsky AS, Thompson BT, Twagirumugabe T, Ware LB, Wick KD. A New Global Definition of Acute Respiratory Distress Syndrome. Am J Respir Crit Care Med. 2024 Jan 1;209(1):37-47. doi: 10.1164/rccm.202303-0558WS. PMID 37487152
- [Result] Habashi NM. Other approaches to open-lung ventilation: airway pressure release ventilation. Crit Care Med. 2005 Mar;33(3 Suppl):S228-40. doi: 10.1097/01.ccm.0000155920.11893.37. PMID 15753733
- [Result] Kucuk MP, Ozturk CE, Ilkaya NK, Kucuk AO, Ergul DF, Ulger F. The effect of preemptive airway pressure release ventilation on patients with high risk for acute respiratory distress syndrome: a randomized controlled trial. Braz J Anesthesiol. 2022 Jan-Feb;72(1):29-36. doi: 10.1016/j.bjane.2021.03.022. Epub 2021 Apr 24. PMID 33905798
- [Result] Borges JB, Okamoto VN, Matos GF, Caramez MP, Arantes PR, Barros F, Souza CE, Victorino JA, Kacmarek RM, Barbas CS, Carvalho CR, Amato MB. Reversibility of lung collapse and hypoxemia in early acute respiratory distress syndrome. Am J Respir Crit Care Med. 2006 Aug 1;174(3):268-78. doi: 10.1164/rccm.200506-976OC. Epub 2006 May 11. PMID 16690982